CLINICAL TRIAL: NCT05823688
Title: Electrical Impedance Tomography (EIT) Monitoring of Regional Ventilation During Pediatric Laparoscopy: an Observational Study
Brief Title: Electrical Impedance Tomography (EIT) Monitoring of Regional Ventilation During Pediatric Laparoscopy
Acronym: Pulmopneumo
Status: Recruiting | Type: Observational
Sponsor: Vittore Buzzi Children's Hospital (Other)
Responsible Party: Principal Investigator, Anna Camporesi, Principal Investigator, Vittore Buzzi Children's Hospital
Other Study IDs: EITPEDLAP
Record Dates: First submitted 2023-04-08; First posted 2023-04-21 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Pediatric Anesthesia; Laparoscopy; Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Electrical Impedance Tomography — Measure of regional ventilation by Electrical Impedance Tomography (EIT) before and during pneumoperitoneum

SUMMARY:
The goal of this prospective, observational study is to describe EIT measurements at different time points during the perioperative period in healthy children undergoing laparoscopic surgery. The objective is to evaluate the impact of general anesthesia and laparoscopy on regional pulmonary ventilation visualized at EIT during the perioperative period.

DETAILED DESCRIPTION:
Electrical impedance tomography (EIT) is a non-invasive, radiation-free functional imaging technique based on image reconstruction of pulmonary regional ventilation by estimating the changes in resistivity (impedance) that occur in the lungs during respiration. Validation data confirms that EIT is highly reproducible and that impedance changes accurately reflect changes in regional ventilation. This allows for the derivation of EIT-derived measurements that can be used to assess bedside regional lung function.

In clinical practice there is increasing emphasis on understanding the impact of anesthesia and mechanical ventilation on regional pulmonary ventilation in order to improve clinical outcomes, including in children.

Several studies have demonstrated that the benefits of using EIT to set ventilatory parameters, improving gas exchange and respiratory mechanics are also applicable outside the intensive care unit. For example, monitoring of changes in regional ventilation in the operating room in adults has been studied to guide intraoperative ventilation setting and adopt it as a strategy to prevent anesthesia-induced atelectasis.

The impact on regional pulmonary ventilation distribution may be significant in situations such as laparoscopic surgery, where capnoperitoneum and Trendelenburg position pose an additional risk of deterioration of respiratory function and may contribute to the development of early postoperative pulmonary complications.In the adult population, studies demonstrate that pneumoperitoneum during laparoscopy can influence the distribution of ventilation together with anesthesia and mechanical ventilation in different ways. In contrast, regional ventilation changes during laparoscopy are still lacking for the pediatric population.

The aim of the present study is to investigate how general anesthesia and capnoperitoneum during laparoscopic procedures can affect the distribution of regional ventilation displayed by EIT in healthy pediatric patients and how these changes correlate with ventilatory parameters and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ASA Status I and II
* elective or urgent laparoscopic procedures (e.g., appendectomy, cholecystectomy, varicocelectomy)

Exclusion Criteria:

* Lack of parental consent
* ASA status III-IV
* Presence of peritonitis or other abdominal inflammatory process that could potentially interfere with spontaneous breathing ventilation
* Need for immediate resuscitation maneuvers
* Severe respiratory illness in the previous 4-6 weeks
* Pre-existing chronic pulmonary conditions
* Concomitant acute pulmonary conditions (e.g. pneumonia, pleural effusion)
* Cardiac arrest
* Skeletal deformities (e.g. rib cage malformations or scoliosis), neuromuscular diseases or cardiac conditions affecting respiratory mechanics
* BMI > 30
* Presence of implantable devices not compatible with EIT (such as pacemakers and implantable defibrillators)

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patients age 10-18 undergoing laparoscopic procedures
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Regional Ventilation distribution | Intraoperative
  Difference in regional ventilation distribution before and after institution of pneumoperitoneum

CONTACTS AND LOCATIONS:
Locations (1):
- Vittore Buzzi Children's Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No